CLINICAL TRIAL: NCT01937416
Title: Safety and Efficacy Investigation of Patients With Diabetic Lower Limb Ischemia by Transplantation of Autologous Bone Marrow Mononuclear Cells
Brief Title: Autologous Bone Marrow Mononuclear Cells Therapy in Diabetic Lower Limb Ischemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Quanhai Li, Director of Cell Thearpy Center, the First Hospital of HeibeiMU, Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12276102D
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes; Lower Limb Ischemia
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- autologous bone marrow mononuclear cells (Experimental): Bone marrow come from the patients himself/herself. With a conventional method and reagent,Ficoll, mononuclear cells were isolated with deleting erythrocyte by density gradient centrifugation.
  Interventions: Biological: autologous bone marrow mononuclear cells

INTERVENTIONS:
Biological: autologous bone marrow mononuclear cells — Bone marrow was taken from patient oneself and mononuclear cells were isolated with deleting erythrocyte by density gradient centrifugation. Bone marrow mononuclear cells were transplanted into ischemia regions of lower limb through intramuscular injection.

SUMMARY:
This study is to evaluate the safety and efficacy of autologous bone marrow mononuclear cells transplantation in diabetic patients with lower limb ischemia.

DETAILED DESCRIPTION:
Diabetic lower limb ischemia as severe complication of diabetes influences the life quality of patients and currently the effective treatment for the disease is lacking. Bone marrow mononuclear cells have been proved to have multiple functions including the differentiation and proliferation. In animal model, bone marrow mononuclear cells could induce angiogenesis and may have therapeutic usage for ischemia disease. The investigators thereby design the study to investigate the possible therapy of diabetic lower limb ischemia with autologous bone marrow mononuclear cells. Patient with diabetic lower limb ischemia was treated with colony stimulating factor for improvement of bone marrow hematopoiesis. Then bone marrow was taken and mononuclear cells were isolated with deleting erythrocyte by density gradient centrifugation. Bone marrow mononuclear cells were transplanted into ischemia regions of lower limb through intramuscular injection. The investigators investigated the safety of the therapy with life signs like temperature, pulse, blood pressure, routine analysis of blood and urine etc. post the transplantation. And the efficacy was evaluated with the measurement of ulcer size, rest pain score, cold sensation score, resting ABI, resting TcPO2, collateral vessel score and skin microcirculation.

ELIGIBILITY:
Inclusion Criteria:

1. fontaine's stage 2-4 or resting ABI <0.7
2. age between 20 and 80 years old
3. sign informed consent, voluntary subjects
4. diagnosis of diabetic lower limb ischemia

Exclusion Criteria:

1. poorly controlled diabetes (HBA1c> 7.0%) and proliferative retinopathy (III-IV stage)
2. malignancy history in the past five years or serum level of tumor markers elevated more than doubled
3. severe heart, liver, kidney, respiratory failure or poor general condition can not tolerate bone marrow mononuclear cells transplantation
4. serious infections (such as cellulitis, osteomyelitis, etc.)
5. pregnant female, or reproductive age female who wants to give birth throughout the course of the study
6. life expectancy less than half a year

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Cell transplantation related side effect | 2 week after cell transplantation
  Temperature,pulse,respiration,blood pressure,routine analysis of blood and urine, liver function,renal function,function of coagulation, ECG,cell transplantation related death and cell transplantation related unexpected amputation

SECONDARY OUTCOMES:
ulcer size | Post cell transplantation: 1, 3, 6 months
  Measuring ulcer area (cm2) and depth (mm)of limb : For each ulcer , photographically record the area and depth with a ruler in order to calculate the ulcer area in square millimeters.
rest pain score | Post cell transplantation: 1,3, 6 months
  Scoring the rest pain based on the degree of pain as following five scales): 0 level-0 point: no pain;
  1. level-1 point: occasional pain which can be recalled;
  2. level-2 points: the pain often but can be tolerated, without or with a little analgesics;
  3. level-3 points: often with need of general analgesics;
  4. level -4 points: affect sleeping due to the pain, general pain medication being difficult to alleviate.
  Before transplantation: points; after transplantation: points.
cold sensation score | Post cell transplantation: 1,3, 6 months
  based on a sense of cold as following five scales: 0 level-0 point: no cold sensation;
  1. level-1 point, or : Occasionally cold feeling;
  2. level-2 points: Often with cold feeling;
  3. level-3 points: significantly cold feeling. and can be significantly improved when using a local insulation.
  4. level-4 points: significantly cold feeling,and can not be significantly improved when using a local insulation.
Resting ABI | Post cell transplantation: 1,3, 6 months
  Measurement of ABI(ankle brachial index, ABI): Measure arterial pressure with a laser Doppler, and then calculate the ankle-brachial index, that is a ratio of ankle arterial blood pressure to brachial arterial blood pressure at rest.
Resting TcPO2 (mmHg) | Post cell transplantation:1, 3, 6 months
  Transcutaneous oxygen pressure(TcPO2) should be measured at the same site in the ischemic limb at rest.
Collateral vessel score | Post cell transplantation: 1,3, 6 months
  Collateral vessel score: Using computed tomographic angiography to score the collateral vessel formation. A mean score is obtained for each ischemic limb by 3 independent interventionists based on the following 4 level score: 0 (no new collateral vessels)
  1. (A little new collateral vessels)
  2. (moderate new collateral blood vessels)
  3. (Rich new collateral vessels)
Skin microcirculation measurement | 1,3,6 months post cell transplantation
  using PeriMed "laser-Doppler flowmetry" measure the skin microcirculation on the same site in the ischemic limb at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Baoyong Yan, Doctor, Study Chair — The First Hospital of Hebei Medical University; Huimin Zhou, doctor, Study Director — The First Hospital of Hebei Medical University; Xu Han, master, Principal Investigator — The First Hospital of Hebei Medical University; Quanhai Li, doctor, Principal Investigator — The First Hospital of Hebei Medical University
Locations (1):
- the First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China